CLINICAL TRIAL: NCT04863898
Title: Improving HIV Treatment Outcomes for People Who Use Drugs: Adapting and Piloting a Drug-use Use Stigma-reduction Intervention in HIV Care and Treatment Clinics in Tanzania
Brief Title: Addressing Drug Use Stigma in Human Immunodeficiency Virus (HIV) Care and Treatment Clinics in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11786; 1R21TW011786-01 (NIH)
Record Dates: First submitted 2021-03-29; First posted 2021-04-28 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Drug Use Stigma in HIV Treatment Clinics
Keywords: Stigma; drug use; people who use drugs; HIV; intervention
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Intervention Model Description: Pilot study to test a drug-use stigma-reduction intervention with staff (study participants) who work in HIV care and treatment clinics. Participants were enrolled, not clinics. This is a single arm study (no comparison group), pre and post survey design with qualitative data collection post pilot intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Staff (Study Participants) Working in HIV Care and Treatment Clinics (Other): Single arm, Pre-post with staff (study participants) working in HIV care and treatment clinics
  Drug use stigma reduction training intervention for staff (study participants) working in HIV care and treatment clinics. The intervention consists of five-2.5 hour participatory training sessions. We will adapt the HP+ health facility HIV stigma-reduction intervention to focus on drug stigma in HIV CTCs. The intervention will address key stigma drivers, including fear, awareness of stigma, and stigmatizing attitudes and beliefs, through a participatory training approach that involves all levels of staff and is grounded in social cognitive theory principles. The approach seeks to reduce stigma through fostering empathy, interpersonal interactions (contact strategies) and building efficacy for stigma reduction through awareness, skills, and knowledge building.
  Interventions: Behavioral: Drug-use stigma reduction intervention for HIV care and treatment clinic staff

INTERVENTIONS:
Behavioral: Drug-use stigma reduction intervention for HIV care and treatment clinic staff — We will adapt the HP+ health facility HIV stigma-reduction intervention to focus on drug stigma in HIV CTCs. The intervention will address key stigma drivers, including fear, awareness of stigma, and stigmatizing attitudes and beliefs, through a participatory training approach that involves all levels of staff and is grounded in social cognitive theory principles. The approach seeks to reduce stigma through fostering empathy, interpersonal interactions (contact strategies) and building efficacy for stigma reduction through awareness, skills, and knowledge building. The intervention consists of five-2.5 hour participatory training sessions.

SUMMARY:
The goal of this study is to adapt and pilot an effective health facility HIV stigma-reduction intervention to address drug use stigma in human immunodeficiency Virus (HIV) Care and Treatment clinics (CTCs) in Tanzania, a barrier to HIV care for People Living with HIV (PLWH) who use drugs. In Tanzania, there are an estimated 300,000 People Who use Drugs (PWUD), primarily heroin. HIV prevalence among PWUD who do not inject (18-25%) and those who do inject (35%) is 4-7 times higher than in the general population (5%). PWUD face high levels of stigma, including when they try to seek HIV treatment at HIV CTCs, presenting a barrier to linkage and retention in HIV treatment for this highly HIV vulnerable group. Reducing drug use stigma in HIV CTCs is critical to improving access to and retention in HIV treatment services for PWUD. In response to this need, the investigators will: 1) Adapt a health facility HIV stigma-reduction participatory training intervention to address drug use stigma in HIV CTCs (Aim 1). 2) Pilot test the adapted drug use stigma-reduction intervention for acceptability, appropriateness, and feasibility (Aim 2).

The investigators will achieve Aim 1 through a systematic, multi-stage adaptation process that will include a formative phase of in-depth interviews with PLWH who use drugs and CTC staff to inform initial adaptation of the Health Policy Plus (HP+) intervention. Stakeholders, including PLWH who use drugs and CTC staff, will provide feedback on the initial materials through a participatory workshop, leading to a training manual that will be reviewed by topic experts and then finalized. Experienced Tanzanian HIV stigma-reduction trainers will deliver the intervention to CTC staff. The pilot test will include 150 staff (the study participants) based in seven CTCs in Dar-es-Salaam. A mixed methods evaluation will comprise pre-post surveys, observation of trainings, and post-training focus group discussions with staff (study participants) who complete the intervention and trainers. Changes in CTC staff (study participants) mean scores on stigma scales from pre- to post-intervention will be assessed, along with measures of intervention acceptability, appropriateness, and feasibility (measured at end line only). Post-intervention focus group discussions will explore themes around the experience of participating in the drug use stigma-reduction training.

DETAILED DESCRIPTION:
The goal of this R21 application is to adapt and pilot an effective health facility human immunodeficiency virus (HIV) stigma reduction intervention to address drug use stigma in HIV CTCs in Tanzania, a barrier to linkage and retention in HIV care PLWH who use drugs. Reducing drug used stigma in HIV CTCs will improve access to and retention in HIV treatment services for PWUD, a key population at elevated risk for HIV, thereby improving individual health outcomes, reducing onward transmission of HIV, and contributing to achievement of the global and national 95-95-95 targets. The investigators propose to do this by adapting (Aim 1) and testing for acceptability, appropriateness and feasibility (Aim 2) a drug use stigma-reduction intervention for HIV CTCs, guided by the eight-step ADAPT-ITT model. The study has two phases. First, the investigators will adapt the participatory training from an evidence-based health facility HIV stigma-reduction intervention (the HP+ total facility approach) to address drug use stigma among HIV CTC staff and then pilot test it with staff (study participants) in seven CTCs in three municipalities of Dar-es-Salaam. The first seven steps of the ADAPT-ITT model will guide AIM 1-the adaptation process, and step eight will guide AIM 2.

Step 1: Assess. Formative research will provide contextual information from PLWH who use drugs and CTC staff, to inform the adaptation of the HP+ intervention to focus on drug use stigma. Given the sensitivity of the topic and concerns about privacy and confidentiality, the investigators will employ individual in-depth interviews with both PLWH who use drugs and CTC staff.

In-depth interviews with PLWH who use opioids: 18 respondents aged 18 or older in the following categories: Medicated Assisted Therapy (MAT) clients living with HIV who get HIV treatment at CTCs; MAT clients not on HIV treatment; PLWH who use opioids who are not on MAT or HIV treatment. With PLWH the investigators will seek to understand the types of drug use stigma (experienced, anticipated, and perceived) that they encounter in relationship to CTCs, the specific manifestations of those types of stigma, and how this stigma influences HIV care linkage and retention among respondents living with HIV. The investigators will also explore what respondents view as driving drug use stigma in CTCs.

In-depth interviews with CTC staff: Fourteen staff from high volume clinics located in areas where people who use drugs congregate or live, who have direct interactions with clients split by type of staff (clinical and non-clinical). The in-depth interviews will focus on capturing stigmatizing attitudes and practices toward PWUD and understanding the underlying drivers of drug use stigma in CTCs (e.g., fear, lack of knowledge, attitudes and beliefs), as well as the who, when, and where drug use stigma occurs in the course of staff-client interactions.

All interviews will be recorded, transcribed, and translated. A multi-stage, modified grounded theory approach to analysis will be deployed, which will include inductive and deductive development of initial codebooks. Coding and analysis will continue iteratively to discover additional themes and issues. The findings will be described in thematic summaries, tables, and diagrams.

Step 2: Decision. Guided by the formative results and the study team's experience working with service delivery for PWUD and developing and adapting stigma-reduction intervention tools for a range of audiences, the study team will conduct the first round of adaptation of the HP+ intervention training curriculum materials. The investigators will develop five, 2.5-hour participatory training modules that can be delivered flexibly across multiple partial days of training. Existing HP+ participatory training modules will be assessed for their appropriateness in terms of training modality (e.g., discussion, role play, reflection) and the specific content that needs to be adjusted (e.g., case studies, pictures, drivers of stigma) to focus on drug use stigma. New materials for identified gaps will be developed, for example, around drug use as a medical condition.

Step 3: Administer. Next, the training materials will be put through a dry run-a 2-day participatory stakeholder workshop with key stakeholders, including HIV CTC staff, people with lived experience of drug use, Community Based Organization staff providing services to PWUD, MAT medical providers, and municipality and ministry of health representatives. Workshop participants will be asked to provide feedback on their overall perceptions and experience of the training (e.g., did it resonate, was it engaging, did it cover the right topics, exercises that should be dropped, gaps that remain to be filled). They will also be asked to comment on the approach and content of each specific exercise, including relevance, appropriateness, and content (including any visual materials).

Step 4: Produce. The study team will review and discuss stakeholder workshop feedback, refining the training manual in response.

Step 5: Topical experts. Two HIV stigma-reduction training experts will review the adapted manual to provide feedback on its congruence with stigma-reduction training principles, the scientific literature, and observed experience of PWUD trying to access HIV treatment.

Step 6: Integrate will involve a final revision of the manual incorporating feedback from the topical experts. Step 7: Trainers, Kimara Peer's two stigma-reduction master trainers and a MAT provider expert and the Principal Investigator (PI) and site PI will work together to finalize training plans.

Step 8: Pilot test. The drug-use stigma-reduction training intervention will be delivered to staff (study participants) in seven HIV CTCs with high client loads located in areas within the three identified municipalities where PWUD congregate or live. These types of CTCs have on average 20 to 25 staff (clinical and non-clinical) who come into direct contact with clients. Staff of all levels will be trained together, which has been shown to have multiple benefits. Training will be on site at the facility and delivered in five, 2.5 hour participatory sessions. Timing of the sessions will be negotiated with each facility to ensure minimal disruption to service delivery, as has been done successfully for the HP+ intervention. Training will be delivered by two master trainers from a local community-based organization (Kimara Peers) who have 20 years of delivering HIV stigma-reduction training, including to health workers, and who also run outreach services and a drop-in center for PWUD and a MAT provider, and an addiction specialist. The training team will include people of lived experience of drug use, who will participate as a panel in one of the sessions.

A mixed-methods approach will be used for assessment: pre-post intervention surveys, training observation, and focus group discussions with CTC staff (study participants) for each cohort of trainees, and one with the intervention trainers. Trainers will complete a process rating form at the end of each session focusing on issues of feasibility, coverage of session content, disruptions, issues raised during the session, and level of participant engagement with the material. The training team will maintain attendance rosters for each session, noting when staff (study participants) leave the room and whether and when they return. The site PI and a member of the field staff will each observe, between them, half of all sessions across the seven facilities, recording observations on the same issues captured by the facilitators, as well as facilitator fidelity to the training manual material and facilitator-participant interaction. Staff (study participants) views on the training will be captured through post-intervention focus groups with 8-12 staff (study participants) who completed the training, one for each cohort of staff trained across clinics. Focus groups will be recorded, transcribed, translated, and analyzed using the same process described above for formative work in Aim 1. Topics will focus on acceptance and appropriateness of training modalities and content, as well as areas where participants wanted more focus. Questions on the length and timing of sessions will also be discussed.

ELIGIBILITY:
Inclusion Criteria:

Intervention pilot testing phase:

-This will include CTC staff and other staff within the medical facility where the CTC is physically housed who come into direct contact with clients attending the CTC (guards, receptionists, lab and pharmacy staff), who work in one of the seven clinics selected for this study.

Exclusion Criteria:

* Under the age of 18.
* Refusal to Consent.
* PLWH participants who appear to be too impaired to provide informed consent or answer questions accurately will be ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura C Nyblade, PhD, Principal Investigator — RTI International
Locations (7):
- Tanzania (7):
  - Amana Hospital, Dar es Salaam
  - Buguruni Health Center, Dar es Salaam
  - Magomeni Health Center, Dar es Salaam
  - Mbagala Kuu, Dar es Salaam
  - Mbagala Rangi Tatu, Dar es Salaam
  - Mnazi Mmoja Hospital, Dar es Salaam
  - Tandale Health Center, Dar es Salaam

IPD SHARING:
Plan to Share IPD: Yes
This 2-year R21 study will adapt and pilot a drug use stigma-reduction intervention for HIV CTCs in Tanzania. The study will produce qualitative data from two phases of the study. In the formative phase, data will include KiSwahili and English transcripts of in-depth interviews with PLWH who use drugs and CTC staff. Qualitative data from the second phase will include focus group discussions with CTC staff who participate in the intervention. The second phase will also include pre-and post-survey data with CTC staff who participate in the intervention. The study investigators are committed to the ideals of collaborative research and resource sharing and are willing to share data and tools developed as part of the proposed research with the broader scientific community. We will provide instruments and protocols, analytic code, and de-identified data to other investigators upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Datasets will be made available after the main findings of the study are accepted for publication.
Access Criteria: Given the sensitive nature of the topic-drug use stigma-being explored in this study, we will make de-identified data and associated documentation available to qualified researchers for non-commercial purposes only under a data sharing agreement that includes commitment to using the data only for research purposes, to securing the data using appropriate computer technology, and to destroying or returning the data after analyses are completed.
  Analytic datasets will be provided as de-identified data files that can be read by common statistical package software, such as SAS or Stata. Electronic codebooks will be provided with all datasets to provide the variable name, label, type, format, positions, consistency codes, and, if applicable, values and value labels.

RESULTS

PARTICIPANT FLOW:
Groups:
- Staff (Study Participants) Working in HIV Care and Treatment Clinics: Pre-post with staff (study participants) working in HIV care and treatment clinics
  Drug-use stigma reduction intervention for staff (study participants) working in HIV care and treatment clinics: We will adapt the HP+ health facility HIV stigma-reduction intervention to focus on drug stigma in HIV CTCs. The intervention will address key stigma drivers, including fear, awareness of stigma, and stigmatizing attitudes and beliefs, through a participatory training approach that involves all levels of staff (study participants) and is grounded in social cognitive theory principles. The approach seeks to reduce stigma through fostering empathy, interpersonal interactions (contact strategies) and building efficacy for stigma reduction through awareness, skills, and knowledge building. The intervention consists of five-2.5 hour participatory training sessions.
Period: Overall Study
Arm/Group | Staff (Study Participants) Working in HIV Care and Treatment Clinics
Started | 151 (This is a single-arm study, pre-post design with staff enrolled (study participants) who work in HIV clinics. Study participants (staff) described here were all placed in the single arm and were offered the intervention. The comparison was pre-post within the single arm for individual participants- (staff)-that is the comparison is before they received the intervention and after they received the intervention. There is no control/comparison arm. Staff were enrolled, not clinics.)
Baseline Survey | 151
Stigma Reduction Intervention | 141 (All study participants (staff) in study were offered stigma-reduction intervention training. For the 10 people who did not receive the training intervention)
Endline Survey | 148 (All participants in study (staff) were requested to complete endline survey, regardless of whether they participated in the stigma-reduction intervention training)
Completed | 141 (141 completed, meaning they both received the stigma-reduction intervention AND completed the endline survey. The outcome measures only include these 141 people in the calculations.)
Not Completed | 10
Not completed — Away from study clinic during intervention training period | 2
Not completed — Preferred not to answer on endline survey why they did not participate in the training | 1
Not completed — Lost to Follow-up | 3
Not completed — Self reported at endline that they had not received information about the training | 1
Not completed — No longer employed at clinic | 3

BASELINE CHARACTERISTICS:
Groups:
- Pre-post With HIV Care and Treatment Clinic Staff: Pre-post with HIV care and treatment clinic staff
  Drug-use stigma reduction intervention for HIV care and treatment clinics: We will adapt the HP+ health facility HIV stigma-reduction intervention to focus on drug stigma in HIV CTCs. The intervention will address key stigma drivers, including fear, awareness of stigma, and stigmatizing attitudes and beliefs, through a participatory training approach that involves all levels of staff and is grounded in social cognitive theory principles. The approach seeks to reduce stigma through fostering empathy, interpersonal interactions (contact strategies) and building efficacy for stigma reduction through awareness, skills, and knowledge building. The intervention consists of five-2.5 hour participatory training sessions.
Arm/Group | Pre-post With HIV Care and Treatment Clinic Staff
Number analyzed (Participants) | 151
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [29 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 151
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — The 7 study clinics where the training took place and at which the staff worked were in the Dar es Salaam region of Tanzania.
  participants
    Tanzania | 151
Highest level of school attended [Number; unit: participants] — This is a categorical variable with the following categories Did not go to school Primary Secondary College/University
  participants
    Did not go to school | 0
    Primary | 32
    Secondary | 40
    College/University | 79
Position in health facility [Count of Participants; unit: Participants]
  Clinical staff | 81
  Non Clinical Staff | 70
Years worked in health facility [Median (Inter-Quartile Range); unit: years] | 4 [3 to 10]
Years worked in HIV care and treatment clinic [Median (Inter-Quartile Range); unit: years] | 4 [2 to 6]
Number of clients treated in past month who use drugs [Median (Inter-Quartile Range); unit: Clients] | 3 [1 to 6.5]
Staff (study participant) count by clinic [Count of Participants; unit: Participants] — This is a count of the number of staff (study participants) in each of the study clinics that participated in this single arm, pre-post study to pilot a drug-use stigma reduction training intervention.
  Participants
    Clinic 1 | 24
    Clinic 2 | 12
    Clinic 3 | 33
    Clinic 4 | 26
    Clinic 5 | 23
    Clinic 6 | 16
    Clinic 7 | 17
Social Desirability Bias [Mean (Standard Deviation); unit: units on a scale] — The Marlowe-Crowne Social Desirability scale (13-items) measures the degree to which a respondent's answers are likely to be influenced by social desirability bias. Each item consists of a dichotomous true/false response, with true indicating that the respondent agrees with the statement. Scores are then calculated by adding together the number of true responses (0 = low degree of social desirability bias; 13 = high degree of social desirability bias). Higher scores correspond to a higher chance that social desirability bias affects the respondent's answers.
  units on a scale | 6.695 (1.999797)
Level of contact with people who use drugs [Count of Participants; unit: Participants] — A 5-item scale that measures the amount that a respondent comes into contact with people who use drugs in professional, social, and personal situations. Each item consists of a dichotomous true/false response, with true indicating that the person agrees with the statement. Scores are calculated dichotomously: agreement with none of the 5 items indicates a low degree of contact ("low contact"), and agreement with one or more of the 5 items indicates a high degree of contact ("high contact").
  Participants
    Low Contact | 48
    High Contact | 103

OUTCOME MEASURES:

1. Primary Outcome: Modified Opening Minds Scale for Health Providers (OMS-HC)
Description: 8-item scale measuring stigma in staff (study participants) working in HIV clinics toward people who use drugs. 5-point Likert scale: 5 indicating the highest degree of agreement with the statement. The score is calculated additively with a range of 8-40. Higher scores indicate a higher level of stigma.
  Included items
  * If I were under treatment for drug addiction, I would not disclose this to any of my colleagues.
  * If I had drug addiction, I would seek treatment at a health facility away from the one I work in.
  * I would see myself as weak if I had drug addiction and could not fix it myself
  * I would be reluctant to seek help if I had drug addiction
  * Despite my professional beliefs, I have negative reactions towards people who use drugs
  * I would not want a person with addiction, even if it were managed, to work with children.
  * Healthcare providers do not need to be advocates for people who use drugs.
  * I am afraid to provide health services to people who use drugs
Time Frame: Baseline survey (weeks 1-3) and Endline Survey (weeks 17-24, 3 months after participant had completed training)
Population: Staff (study participants) who completed the training intervention and answered all of the component questions of the OMS scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff (Study Participants) Working in HIV Care and Treatment Clinics
Number analyzed (Participants) | 132
score on a scale
  Baseline | 22.92 (4.78)
  Endline | 16.82 (4.02)
Statistical Analysis 1: Comparison: Staff (Study Participants) Working in HIV Care and Treatment Clinics; Using the PASS software program, we estimated the power for comparisons of scores from pre- to post-intervention, assuming a p-value of 0.05 (two-sided) and a final sample size of 131 with both measurements. We would have 85% power to detect a small-to-medium sized effect based on standardized mean difference (d=0.32); Test type: Superiority; Mean Difference (Net) = -6.1, 95% CI 2-sided [-7 to -5.2] — LME regression, random intercepts by individual and fixed effects of participant characteristics. Difference = endline - baseline

2. Primary Outcome: Feasibility of Intervention Measure
Description: A 4-item scale that measures staff's (study participants') perception of the feasibility of the intervention in their context. Each item consists of a 5-point Likert scale, with 5 indicating the highest degree of agreement with the item. The score is calculated by taking the mean of the responses. Scores range from 1-5. Higher values correspond to a higher degree of agreement that the intervention is feasible in the respondent's context.. The questions are:
  1. (INSERT INTERVENTION) seems implementable.
  2. (INSERT INTERVENTION) seems possible.
  3. (INSERT INTERVENTION) seems doable.
  4. (INSERT INTERVENTION) seems easy to use.
Time Frame: Endline Survey (weeks 17-24, 3 months after participant had completed training)
Population: Clinic Staff who were participants in the study who completed the training intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff (Study Participants) Working in HIV Care and Treatment Clinics
Number analyzed (Participants) | 141
score on a scale | 4.7 (0.33)

3. Primary Outcome: Acceptability of Intervention Measure
Description: A 4-item scale that measures the degree to which staff (study participants) find the intervention acceptable. Each item consists of a 5-point Likert scale, with 5 indicating the highest degree of agreement with the item. The score is calculated by taking the mean of the responses. Scores range from 1-5. Higher values correspond to a higher degree of agreement that the intervention is acceptable to the respondent. The questions are:
  1. (INSERT INTERVENTION) meets my approval.
  2. (INSERT INTERVENTION) is appealing to me.
  3. I like (INSERT INTERVENTION).
  4. I welcome (INSERT INTERVENTION).
Time Frame: Endline Survey (weeks 17-24, 3 months after participant had completed training)
Population: Participants who completed the training intervention
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Staff (Study Participants) Working in HIV Care and Treatment Clinics
Number analyzed (Participants) | 141
score on a scale | 4.72 (0.35)

4. Primary Outcome: Appropriateness of Intervention Measure
Description: A 4-item scale that measures the degree to which staff (study participants) find the intervention acceptable. Each item consists of a 5-point Likert scale, with 5 indicating the highest degree of agreement with the item. The score is calculated by taking the mean of the responses. Scores range from 1-5. Higher values correspond to a higher degree of agreement that the intervention is acceptable to the respondent. The questions are:
  1. (INSERT INTERVENTION) seems fitting.
  2. (INSERT INTERVENTION) seems suitable.
  3. (INSERT INTERVENTION) seems applicable.
  4. (INSERT INTERVENTION) seems like a good match.
Time Frame: Endline Survey (weeks 17-24, 3 months after participant had completed training)
Population: Participants who completed the training intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Staff (Study Participants) Working in HIV Care and Treatment Clinics
Number analyzed (Participants) | 141
score on a scale | 4.82 (0.33)

5. Secondary Outcome: Knowledge About Drug Use and How to Provide HIV Services to People Who Use Drugs
Description: Self-reported knowledge. Likert scale (1-5): 8-10 items (2 additional items for clinical staff (CS)). Scores (range:1-5), calculated by taking the mean value of responses to all questions. Higher scores correspond to higher degrees of knowledge and therefore a better outcome.
  Items
  * I feel
    * I have a working knowledge of drugs and drug related problems.
    * safe providing HIV services to people who use drugs (PWUD)
  * I feel I know enough about {insert below item} to carry out my role providing HIV services to PWUD
    * the causes of drug problems
    * the physical effects of drug use
    * the psychological effects of drugs
    * the factors which put people at risk of developing drug problems
  * I feel I know enough about {insert below item} to provide appropriate services to PWUD
    * drug addiction as a brain disease
    * the social effects of drug use
    * drug-to drug interactions (CS only)
    * co-occurring conditions (CS only)
Time Frame: Baseline survey (weeks 1-3) and Endline Survey (weeks 17-24, 3 months after participant had completed training)
Population: Participants who completed the training intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pre-post With HIV Care and Treatment Clinic Staff
Number analyzed (Participants) | 141
score on a scale
  Baseline | 3.4 (0.71)
  Endline | 4.37 (0.49)
Statistical Analysis 1: Comparison: Pre-post With HIV Care and Treatment Clinic Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.97, 95% CI 2-sided [0.86 to 1.09] — Calculated using a linear mixed effect regression model with random intercepts by individual Difference = endline - baseline

6. Secondary Outcome: Modified Bogardus Social Distance Scale
Description: 6-item scale measuring social distance, or (un)willingness to interact with a person who uses drugs in different social interactions. 4-point Likert scale, with 4 indicating a response of "definitely yes" and 1 indicating "definitely no". The score is calculated additively with a range of 6-24. Higher scores correspond to higher degrees of social distance and therefore a worse outcome.
  Included items
  * Would you feel ashamed if people knew someone in your family has drug addiction?
  * Would you be afraid to have a conversation with someone who uses drugs?
  * Would you be disturbed about working at the same health facility with someone who uses drugs?
  * Would you stop being friends with someone who uses drugs?
  * Would you feel upset or disturbed being in the same room with someone who uses drugs?
  * Would you marry someone who uses drugs? (reverse coded)
Time Frame: Baseline survey (weeks 1-3) and Endline Survey (weeks 17-24, 3 months after participant had completed training)
Population: Participants who completed the training intervention and answered all of the component questions of the Modified Bogardus Social Distance Scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pre-post With HIV Care and Treatment Clinic Staff
Number analyzed (Participants) | 141
score on a scale
  Baseline | 12.6 (3.16)
  Endline | 8.34 (2.07)
Statistical Analysis 1: Comparison: Pre-post With HIV Care and Treatment Clinic Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -4.2, 95% CI 2-sided [-4.7 to -3.6] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: No data was collected as this was a pilot study of a stigma-reduction training intervention with HIV care and treatment clinic staff (participants) and does not involve any physical or biological change. The only risk to participants (clinic staff participating in the training) is social discomfort with the topic area they are receiving training in (stigma).
Description: This particular intervention, which was pilot testing a stigma-reduction training intervention with HIV care and treatment clinic staff (participants), does not involve any physical or biological change. The only risk to participants (clinic staff participating in the training) is social discomfort with the topic area they are receiving training in (stigma).
Arm/Group | Staff (Study Participants) Working in HIV Care and Treatment Clinics
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT04863898/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT04863898/SAP_001.pdf